CLINICAL TRIAL: NCT03649490
Title: A Prospective Multicenter Study Evaluating the Effect of Implant Material and/or Surface Structure on Progression of Fusion in XLIF® Surgery
Brief Title: Advanced Materials Science in XLIF Study
Acronym: AMS in XLIF
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.X1801
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Smooth PEEK Interbody Implants in XLIF: Smooth PEEK interbody implants for XLIF (with allograft chips and BMA or cancellous allograft) provide maximum surface area and structural stability with large central apertures to allow bony through-growth. Multiple length options enable optimal apophyseal support, thus reducing the chance of subsidence. Additionally, lordotic profiles are available to induce proper sagittal alignment.
- 3D-Printed Titanium Interbody Implants in XLIF: 3D-printed, fully porous titanium interbody implants for XLIF (with allograft chips and BMA or cancellous allograft) have a porous architecture that mimics the porosity and stiffness of bone for reduced stress shielding and improved radiographic imaging. The advanced microporous surface topography creates an ideal environment for bone in-growth.
- Porous PEEK Interbody Implants in XLIF: Porous PEEK interbody implants for XLIF (with allograft chips and BMA or cancellous allograft) combine the osseointegration capabilities of porous metal implants with the favorable imaging and mechanical properties of traditional PEEK implants. The Porous PEEK architecture, with 60% porosity and 300 mm average pore size, is specifically tailored to elicit the optimal osteogenic cell response and promote bone tissue ingrowth inside the pores, as demonstrated in preclinical studies.

SUMMARY:
This study is being conducted to evaluate the clinical and radiographic outcomes of three different interbody implant types when used with cancellous allograft chips with BMA or cellular allograft in patients undergoing XLIF surgery. The study will evaluate success by comparing the rate of fusion, complications profile, and any relationships between clinical outcomes (pain and function) and radiographic outcomes (fusion rate) between the three implant groups.

DETAILED DESCRIPTION:
This study is a prospective, non-concurrent, multicenter study to compare the clinical and radiographic outcomes of smooth PEEK, 3D-printed titanium, and Porous PEEK interbody implants when used with cancellous allograft chips with BMA or cellular allograft in subjects who undergo XLIF surgery at one or two levels. To minimize selection bias, all consecutive patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. These patients will present with degenerative conditions in the lumbar spine that are amenable to surgical treatment and will be screened prior to study enrollment. Once enrolled into the study, subjects will undergo their XLIF operation using one of the 3 previously noted interbody implants based on a non-concurrent enrollment schedule. The bone graft material used inside the interbody implant will be randomly assigned between cancellous allograft chips with BMA or cellular allograft prior to surgery based on surgeon investigators' equipoise for the effectiveness of both bone graft materials. Subjects will be followed for 24 months following surgery to determine the number of study subjects that are solidly fused at or before 24 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who are 18-80 years of age;
2. Planned interbody fusion surgery, including at least one level of extreme lateral interbody fusion (XLIF) prior to enrollment in the research at one or two consecutive lumbar levels for degenerative disc disease, including those with up to Grade 2 spondylolisthesis, with one of the following NuVasive, Inc. interbody implants:

   1. Coroent® XL PEEK interbody implant; or
   2. Modulus® 3D-printed titanium interbody implant; or
   3. Cohere® XLIF Porous PEEKTM interbody implant.

   If a transforaminal lumbar interbody fusion or anterior lumbar interbody fusion (TLIF or ALIF) is planned adjacent to the XLIF level, the same NuVasive, Inc. interbody implant material type must be used as determined by the implant enrollment schedule. For example:
   1. Smooth PEEK: Coroent XL PEEK (XLIF) + Coroent L (TLIF) or Coroent XLR (ALIF) or Brigade (ALIF)
   2. 3D-printed titanium: Modulus XLIF + Modulus TLIF or Modulus ALIF
   3. Porous PEEK: Cohere XLIF + Coalesce TLIF (currently no ALIF option)
3. The planned procedure must include placement of bilateral posterior screw fixation with or without intrafacet fusion using autograft (with or without the assigned allograft used at the XLIF level(s)) at the treated level(s). Direct posterior decompression at the index interbody fusion level(s) is acceptable.
4. Preoperative coronal Cobb angle of < 10°;
5. Able to undergo surgery based on physical exam, medical history, and surgeon judgment;
6. Understands the conditions of enrollment and willing to sign an informed consent to participate in the evaluation.

Exclusion Criteria:

1. Use of BMP, synthetic bone graft substitutes, allografts, or any other graft material in the interbody or intrafacet spaces other than those under study;
2. Posterior grafting other than the allowed intrafacet fusion at the treated level(s);
3. Revision of prior fusion at treated level(s) (adjacent level interbody fusion is acceptable);
4. XLIF procedure that requires or results in the release of the anterior longitudinal ligament or posterior osteotomy;
5. Preoperative coronal Cobb angle of ≥ 10°;
6. Procedures performed with XLIF interbody implants with integrated vertebral body screw(s);
7. Active smoking six (6) weeks prior to surgery;
8. Systemic or local infection (active or latent);
9. Diseases that significantly inhibit bone healing (e.g., prior diagnosis of osteoporosis, metabolic bone disease, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease);
10. Rheumatoid arthritis or other autoimmune disease that, in the option of the investigator, would interfere with bone healing and/or fusion;
11. Treatment with pharmaceuticals interfering with calcium metabolism;
12. Undergoing chemotherapy or radiation treatment or chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery or anytime postoperatively, other than episodic use or inhaled corticosteroids);
13. Use of bone stimulators postoperatively;
14. Non-ambulatory, wheelchair-bound;
15. Involvement in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested);
16. Significant general illness (e.g., HIV, active metastatic cancer of any type, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease);
17. Spinal metastases or active spinal tumor malignancy;
18. Immunocompromised or is being treated with immunosuppressive agents;
19. Pregnant, or plans to become pregnant during the study;
20. Mental or physical condition that would limit the ability to comply with study requirements;
21. Prisoners;
22. Participating in another clinical study that would confound study data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who are 18-80 years of age with planned extreme lateral interbody fusion (XLIF) surgery prior to enrollment in the research at one or two lumbar levels for the treatment of degenerative disc disease, including those with up to Grade 2 spondylolisthesis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion Success | 24 months
  The proportion of subjects with apparent radiographic fusion at or before 24 months within each treatment group

SECONDARY OUTCOMES:
MCID and SCB threshold for each PRO: VAS (back/leg pain), ODI, and EQ-5D, within each treatment group | 3, 6, 12, and 24 months
  Percentage of subjects meeting minimal clinically important difference (MCID) and substantial clinical benefit (SCB) thresholds for each patient-reported outcome (PRO): Back and leg pain (visual analog scale (VAS)), disability (Oswestry disability index (ODI)), and quality of life (EQ-5D) within each treatment group.
Fusion Rates at Follow-up Timepoints | 6, 12, 24 months
  Percentage of subjects with a successful radiographic interbody fusion by each follow-up timepoint (6, 12, and 24-month postoperative follow-up)
Maintenance of Radiographic Correction | 3, 6, 12, and 24 months
  Percentage of subjects with maintenance of radiographic correction out to 24-months postoperative follow-up within each treatment group
Complications | 3, 6, 12, and 24 months
  Rate of complications attributable to the use of the interbody implants to be studied

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — Globus Medical
Locations (15):
- United States (15):
  - Hartford Healthcare Bone and Joint Institute, Hartford, Connecticut
  - Lyerly Neurosurgery, Jacksonville, Florida
  - University of South Florida Department of Neurosurgery, Tampa General Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Suburban Hospital, Johns Hopkins Medicine, Bethesda, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia Orthopedic Group Research, Columbia, Missouri
  - OrthoCarolina, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Atlantic Brain and Spine, Wilmington, North Carolina
  - The Spine Clinic of OKC, Oklahoma City, Oklahoma
  - UT Health San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Evergreen Health, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No